CLINICAL TRIAL: NCT06010498
Title: The Effect of Eye Mask Applied on Patients Undergoing Coronary Artery Bypass Graft Surgery on Sleep Quality and Pain: Double-Blind Randomized Controlled Study
Brief Title: The Effect of Eye Mask Applied on Patients Undergoing Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Necibe Dağcan, Lecturer, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KutahyaHSU-NECIBE-DAGCAN-0002
Record Dates: First submitted 2023-08-11; First posted 2023-08-24 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Sleep Disorder; Pain, Postoperative
Keywords: Heart Surgery; pain; CABG; eye mask; nursing; sleep quality; randomized controlled trial
MeSH Terms: conditions — Coronary Artery Disease; Sleep Wake Disorders; Pain, Postoperative; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Mask Group (Experimental)
  Interventions: Behavioral: eye mask; Behavioral: standart care
- Standart Care (No Intervention)

INTERVENTIONS:
Behavioral: eye mask — * First day morning The Introductory Characteristics Form will be filled.
  * First day night Standard care will be given
  * Second day morning Richards-Campbell Sleep Questionnaire and Numerical Pain Scale to be filled
  * Second day night Standard care will be given + eye patch will be applied (22:00-06:00)
  * Third day morning Richards-Campbell Sleep Questionnaire and Numerical Pain Scale to be filled
  * Third day night Standard care will be given + eye patch will be applied (22:00-06:00)
  * Fourth day morning Richards-Campbell Sleep Questionnaire and Numerical Pain Scale to be filled
  Arms: Eye Mask Group
Behavioral: standart care — Control group (n)
  * First day morning The Introductory Characteristics Form will be filled.
  * First day night Standard care will be given
  * Second day morning Richards-Campbell Sleep Questionnaire and Numerical Pain Scale to be filled
  * Second day night Standard care will be given
  * Third day morning Richards-Campbell Sleep Questionnaire and Numerical Pain Scale to be filled
  * Third day night Standard care will be given)
  * Fourth day morning Richards-Campbell Sleep Questionnaire and Numerical Pain Scale to be filled
  Arms: Eye Mask Group

SUMMARY:
Introduction: Coronary Artery Bypass Graft (CABG) performed with open heart surgery technique is a successful operation in the treatment of cardiovascular diseases. Incision of the sternum region, saphenous vein graft, sternal retraction, presence of chest and mediastinal tubes cause pain. The pain experienced by the patients, the complications related to the disease they have, and the stress they experience cause an increase in sleep problems. In addition, the increase in sympathetic activity after surgery and nursing care interventions also affect sleep quality. The literature reports that sleep disorders affect the working physiology of the heart in patients with cardiac disease, adversely affect heart health and affect postoperative recovery. In addition, since sleep disorders are also associated with cardiovascular diseases, it is of great importance to improve the sleep quality of this group of patients. One of the non-pharmacological nursing interventions is the eye patch. The eye patch is an instrument made of fabric, with an elastic strap, aimed at pure darkness by diverting all light from the patient's eyes. The main physiological purpose of using an eye patch is to adjust the hormones melatonin and cortisol, which affect the circadian rhythm. As a result, it is thought that the eye patch will prevent patients from being exposed to excessive light in the hospital environment, the regulation of hormones and sleep quality will improve, and the pain will decrease.

Purpose: The aim of this study is to examine the effect of eye patch applied to patients undergoing coronary artery bypass graft surgery on sleep quality and pain.

Method: Individuals who have undergone coronary artery bypass graft surgery in accordance with the sampling inclusion criteria will be randomly assigned to the experimental and control groups by block randomization. After determining the groups, each patient in the experimental and control groups, whose written consent was obtained, will have the first researcher fill out the Descriptive Characteristics Form, Richards-Campbell Sleep Questionnaire and Numerical Pain Scale on the morning of the first night they spent in the clinic.

Patients in the experimental group will be given the "standard care" and "eye patch" application in the clinic on their 2nd and 3rd nights in the clinic. The patients in the control group will only be provided with the "standard care" in the clinic on their 2nd and 3rd nights in the clinic. Patients in both groups will be asked to fill out the Richards-Campbell Sleep Questionnaire and Numerical Pain Scale forms in the mornings of the 2nd and 3rd nights.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) are among the leading causes of death globally. Coronary Erter Bypass Graft (CABG) performed with open heart surgery technique is a successful operation in the treatment of cardiovascular diseases. In the face of this life-threatening experience, patients face many stressors until discharge, and pain is one of them and causes anxiety. Incision of the sternum region, saphenous vein graft, sternal retraction, presence of chest and mediastinal tubes cause pain. Mild to moderate pain persisting until the post-operative 7th day indicates that pain persists as an important postoperative problem in this patient group. The pain experienced by the patients, the complications related to the disease they have, and the stress they experience cause an increase in sleep problems. In addition, the increase in sympathetic activity and nursing care interventions after surgery also affect sleep quality.Nurses are responsible for meeting the basic life needs of the patients they care for. The most important of these needs is sleep. Sleep deprivation causes cognitive problems in patients, affects the immune system, and causes nosocomial infections, affecting recovery time. The literature reports that sleep disorders affect the working physiology of the heart in patients with cardiac disease, adversely affect heart health and affect postoperative recovery. In addition, deterioration of sleep quality causes more pain and increased pain intensity, delaying wound healing. In addition, since sleep disorders are also associated with cardiovascular diseases, it is of great importance to increase the sleep quality of this group of patients. There are many factors that affect the sleep quality of patients. The most important factor that impairs sleep quality is light. Inexpensive and non-pharmaceutical methods can be preferred to improve the sleep quality of patients. Environmental regulations can improve sleep quality. Therefore, it is reported that environmental changes such as dim and dark clinics increase sleep quality. Apart from these, one of the non-pharmacological nursing interventions is the eye patch. The eye patch is an instrument made of fabric, with an elastic strap, aiming at pure darkness by diverting all light from the patient's eyes.The main physiological purpose of using an eye patch is to adjust the hormones melatonin and cortisol, which affect the circadian rhythm. As a result, it is thought that the eye patch will prevent patients from being exposed to excessive light in the hospital environment, the regulation of hormones and sleep quality will improve, and the pain will decrease. There are many studies in the literature on the sleep quality of patients using eye patches, and the results show that the eye patch improves sleep quality. However, from a limited number of studies examining the effects of eye patch on sleep and pain in patients who have undergone cardiac surgery. Due to the limited number of studies, it was aimed to examine the effect of eye patch applied to patients undergoing coronary artery bypass graft surgery on sleep quality and pain.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Those under 65 (Studies show that nighttime awakenings and sleep durations change with age (Lie et al., 2018)
* Can speak Turkish
* Those who agreed to participate in the study
* Those who have not had open heart surgery before
* No emergency bypass surgery
* No intra-aortic balloon pump or pacemaker
* Not taking inotropic drugs
* Those who have not consumed coffee or hypnotic drugs at least 12 hours before
* Those who have not been working the night shift for the last 3 months
* No history of chronic pain (eg arthritis)
* Able to wear an eye mask on their own
* Not addicted to alcohol and drugs
* Does not have a psychological problem (such as depression, anxiety disorder)
* No anxiolytic use
* No chronic sleep problems
* Not using sleeping pills

Exclusion Criteria:

* Low risk factor for complications (eg ejection fraction < 35%).
* During CABG surgery, mitral valve repair or replacement (Each type of heart surgery will differ in terms of operation time, site of surgery, recovery time, and length of hospital stay, which may affect the patient's anxiety.)
* Patients with chest tube and drain
* Patients with vision problems
* Patients with hearing problems
* Patients with claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
sleep quality measurement (Richards- Campbell Sleep Questionnaire) | Once a day on the second day in the morning, on the third day in the morning, on the fourth day in the morning
  Richards- Campbell Sleep Questionnaire: Developed by Richards in 1987, the Richard-Campbell Sleep Questionnaire (RCSQ) is a 6-item scale that evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart between 0 and 100 with the visual analog scale technique. A score of "0-25" from the scale indicates very bad sleep, and a score of "76-100" indicates very good sleep. As the score of the scale increases, the sleep quality of the patients also increases. The Cronbach α value of the scale developed by Richards was found to be 0.82. The Turkish validity and reliability of the scale was investigated by Özlü and Özer in 2015 and the Cronbach α value was found to be 0.91.
pain measurement (numerical pain scale) | Once a day on the second day in the morning, on the third day in the morning, on the fourth day in the morning
  Numerical Pain Scale:It is based on the expression of pain intensity in numbers. While the absence of pain is expressed as 0 in numerical scales, the number shown increases as the severity of pain increases, and 10 points represent unbearable pain. Numerical scales have been adopted more because they facilitate the definition of pain severity and facilitate scoring and recording.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu NAL, Msc RN, Principal Investigator — kütahya health sciences university; Gülşah GÜROL ARSLAN, Msc RN, Principal Investigator — Dokuz Eylul University; Mehmet Ali ASTARCIOĞLU, Doctor, Principal Investigator — kütahya health sciences university; Ali İhsan PARLAR, Doctor, Principal Investigator — kütahya health sciences university; Necibe DAĞCAN, Msc RN, Principal Investigator — Dokuz Eylul University
Locations (1):
- Necibe, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided